CLINICAL TRIAL: NCT03779568
Title: Determination of ED50 and ED95 of Isobaric Bupivacaine for Post-Partum Bilateral Tubal Ligation
Brief Title: ED50 and ED95 of Isobaric Bupivacaine for Post-Partum Bilateral Tubal Ligation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU 082018-026
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose adjustment of bupivacaine (Experimental): Patient will receive isobaric bupivacaine based on previous patient experience.
  Interventions: Other: Dose adjustment of bupivacaine

INTERVENTIONS:
Other: Dose adjustment of bupivacaine — Spinal bupivacaine dose will be adjusted according to previous patient experience.
  Other Names: Spinal bupivacaine dose adjustment

SUMMARY:
Spinal anesthesia is one of the preferred anesthetic techniques for post-partum bilateral tubal ligation (PBTL). Bupivacaine is the most commonly used local anesthetic for neuraxial anesthesia for post-partum tubal ligation. Typically, hyperbaric bupivacaine would be injected into the spinal (intrathecal) space via a spinal needle; however, ongoing medication shortages have resulted in limited availability on a local and national level. One proposed alternative is isobaric bupivacaine; however, studies investigating its use for post-partum bilateral tubal ligation are limited.

The purpose of this prospective study is to determine the minimal effective dose (ED50 and ED95) of isobaric bupivacaine for adequate anesthesia during post-partum tubal ligation after vaginal delivery.

DETAILED DESCRIPTION:
This prospective study proposes to enroll 40 post-partum women who are undergoing elective post-partum bilateral tubal ligation. The patient will be positioned sitting, and combined spinal anesthesia will be performed at L2-3 or L3-4 level. The presence of an epidural catheter enables the provider to supplement the spinal anesthetic if required. The starting dose of isobaric bupivacaine will be 10 mg based on prior similar studies1,4 and our institution's current practice. The dose of intrathecal isobaric bupivacaine was decided by using the up-down sequential method.

The motor block will be graded by a modified Bromage score: Score 1 = complete block, unable to move feet or knees; 2 = almost complete block, able to move feet only; 3 = partial block, just able to move knees; 4 = detectable weakness of hip flexion while supine, full flexion of knees; 5 = no detectable weakness of hip flexion while supine; and 6 = able to perform partial knee bend. The score of 1 or 2 within 10-15 minutes of injection will be evaluated as successful motor block.

The success of the sensory spinal block will be noted when bilateral T6 sensory level to pinprick is attained after 10 mins from the intrathecal drug administration, this is in accordance with previous studies1.

If spinal anesthesia is inadequate, the epidural catheter will be dosed up for supplementation. All observations, including block characteristics and the associated outcome (i.e., adequate or inadequate block), will be evaluated by a dedicated anesthesia provider.

Intraoperative adverse effects, such as hypotension, bradycardia, nausea, or vomiting, pruritus, or shivering were noted. Hypotension is defined as a decrease of more than 20% in basal systolic blood pressure within 30 minutes of intrathecal injection. The management of blood pressure including dose of pressor: phenylephrine and ephedrine will be at the discretion of the attending anesthesiologist. The use of pressor and anti-emetics will also be recorded.

The study will be take place in standard clinical context. The study does not deviate from our current practice, which includes the use of combined spinal anesthesia where the epidural catheter is available if supplemental local anesthetic is required.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Patients undergoing elective post-partum bilateral tubal ligation after vaginal delivery
* Patients receiving spinal epidural anesthesia with combination of bupivacaine and fentanyl

Exclusion Criteria:

* American Society of Anesthesiologists physical status score >3,
* Contraindications to neuraxial analgesia
* Patients in whom a combined spinal epidural cannot be performed
* Body mass index >40 kg/m2
* Allergy or hypersensitivity to local anesthetics and fentanyl
* Severe liver, kidney or respiratory disease.
* Inability to understand the study protocol
* Refusal to provide written consent

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2020-04-09 (Actual)

PRIMARY OUTCOMES:
Success or failure of the intrathecal block | Perioperative
  The score of 1 or 2 within 10-15 minutes of injection will be evaluated as successful motor block.

CONTACTS AND LOCATIONS:
Overall Officials: Seema Dave, MPH, Study Chair — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No